CLINICAL TRIAL: NCT02213419
Title: EUS-guided Double Ethanol Lavage for Pancreatic Cysts: a Prospective Cohort Study
Brief Title: Endoscopic Ultrasonography-guided Double Ethanol Lavage for Pancreatic Cysts: a Prospective Cohort Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-06-058-001
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2014-07

CONDITIONS: Pancreatic Mucinous-Cystic Neoplasm
Keywords: Cystic Tumors of the Pancreas; Endoscopic Ultrasound; Ethanol
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ethanol double lavage (Experimental): Endoscopic ultrasonography-guided double ethanol lavage
  Interventions: Drug: Endoscopic ultrasonography-guided double ethanol lavage

INTERVENTIONS:
Drug: Endoscopic ultrasonography-guided double ethanol lavage — A radial echoendoscope and a 22 gauge needle were then used for cyst fluid aspiration and ethanol lavage.
  The 80 percent volume of cyst fluid was aspirated, and the pure ethanol was injected into the collapsed cyst until the original shape was restored. After 3-5 minutes, the reaspiration of the injected ethanol was then performed. The pure ethanol was reinjected into the collapsed cyst, followed by reaspiration of maximal possible volume for 3-5 minutes.
  Other Names: Ethanol

SUMMARY:
Due to widespread use of cross-sectional imaging modalities, pancreatic cysts are common in abdominal image. These lesions encompass a wide spectrum, ranging from benign to malignant. The diagnosing specific type of cystic lesion is limited in spite of recent advances of diagnostic modalities. Surgical resection is generally recommended for malignant and potentially malignant lesions. However, surgical resection has significant morbidity and sometimes mortality. Recently, a few study of EUS-guided ethanol lavage for cystic tumors of the pancreas reported that complete resolution was achieved in only one-third of patients. Ethanol lavage of pancreatic cysts may be alternative method to surgical resection.

The purpose of this study is the double ethanol lavage is a safe and effective method for treatment in those with the indeterminate pancreas cysts.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older of any gender, ethnicity and race
* Voluntary enrollment and ability to give written informed consent
* Capable of safely undergoing endoscopy with deep sedation or general anesthesia
* Indeterminate cystic lesion which was diagnosed in cross-sectional image (CT and MRI)
* Pancreatic cystic lesion having uni- or oligo-locular (defined as having 2-6 locules within a cyst) and 2~4 cm in diameter

Exclusion Criteria:

* Pancreatic cystic lesions which had the typical morphology of serous cystadenomas (i.e., honeycomb appearance) and pseudocysts (i.e., recent history of acute pancreatitis or parenchymal changes)
* Pancreatic cystic lesions having communication between the cystic lesion and the main pancreatic duct according to endoscopic retrograde cholangiopancreatography and magnetic resonance cholangiopancreatography
* Pancreatic cystic lesions having overt evidence of carcinomas, such as peripancreatic invasion
* Patients with a bleeding tendency (prothrombin time > 1.5 international normalized ratio [INR] or platelet count < 50,000/μL).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Subjects with Complete or Partial response of treatment | 1 year after final treatment
  Complete or partial response of treatment will be defined by the presence of a treated cystic structure, and its volume and maximum diameter in cross-sectional imaging studies (CT, MR)

SECONDARY OUTCOMES:
Incidence rate of adverse events after treatment | 1 year after final treatment
  Adverse events include pancreatitis, bleeding, perforation, any other occurrence resulting in hospitalization, medical treatment, surgery, death, or disability

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Kyun Lee, M.D., Ph.D., Principal Investigator — Division of Gastroenterology, Samsung Medical Center
Locations (1):
- Samsung Medical Cencer, Seoul, South Korea